CLINICAL TRIAL: NCT04637945
Title: a Randomized Placebo-controlled Study Investigating the Effects of a Long-term Dietary Supplementation With an Anthocyanin-rich Blend on the Metabolic and Inflammatory Responses to a High-fat Meal in Healthy Subjects
Brief Title: Inflammatory and Metabolic Responses to Long-term Dietary Supplementation With Anthocyanin-rich Blend
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pharmanex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20-PHX-0002
Record Dates: First submitted 2020-08-05; First posted 2020-11-20 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Anthocyanins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): The placebo will be delivered in softgels consisting of colorant, olive oil, sunflower lecithin, yellow beeswax, bovine gelatin, glycerin and water.
  Interventions: Other: Placebo
- ACRB (Experimental): The ACRB product will be delivered in softgels consisting of anthocyanin-rich blend. Each softgel will contain: i) 49 mg bilberry extract; ii) 101 mg black currant extract; and iii) 303 mg black rice extract. The high ACRB will deliver at least 108 mg anthocyanins. The product will also contain olive oil, sunflower lecithin, yellow beeswax, bovine gelatin, and water.
  Interventions: Dietary Supplement: ACRB

INTERVENTIONS:
Dietary Supplement: ACRB — Product will be consumed once daily, preferably with breakfast.
  Arms: ACRB
Other: Placebo — Product will be consumed once daily, preferably with breakfast.
  Arms: placebo

SUMMARY:
This study will investigate the capacity of an anthocyanin-rich blend (ACRB) dietary supplement to improve the alterations in lipid and glucose homeostasis triggered by consumption of a high-fat meal. Given the impact of Western style diets and obesity on the development of type 2 diabetes, cardiovascular disease and other pathologies, this study has major public health implications.

DETAILED DESCRIPTION:
In particular, this study will investigate the beneficial effects of long-term (8 weeks) supplementation with ACRB on fasting and postprandial levels of plasma triglycerides, as well as other parameters of lipid and glucose homeostasis and inflammation. Postprandial changes will be evaluated after consumption of a high-fat meal.

Subjects will receive either a: i) placebo (control),or ii) ACRB product for 8 weeks. At the beginning and at the end of the 8-week period, subjects will be submitted to a metabolic challenge consisting of consuming a high-fat meal after receiving the study product (placebo, ACRB). The high-fat meal will consist of English muffin bread, sausage, egg and cheese, obtained from US market with carotenoid-free palm oil added to bring the total dietary fat to the desired level. The total weight of the high-fat meal will be 320 g with 70.5 g of fat (29.8 g of saturated fat), 270 mg of cholesterol, 65 g carbohydrate, 5.2 g sugar, and 33 g protein. The total energy content of the high-fat meal will be 1,026 Kcal with a total of 62% energy originated from fat, 25% from carbohydrates and 13% from protein. Blood will be taken by venipuncture before (baseline, 0 h) and 0.25, 0.5, 1, 2, 3 and 5 h after consumption of both the high-fat meal and the study product. Plasma will be collected and chylomicrons and peripheral blood monocytes (PBMCs) will be isolated. Blood pressure and skin carotenoid content will be measured. Subjects will be also asked to collect feces before starting and at the end of the 8 week period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is healthy and, in the opinion of the investigator, free of any medical conditions that might affect study measurements.
2. Male or female.
3. Age between 18 - 40 years inclusive.
4. BMI between 21 - 29.9 kg/m2.
5. Female subject of childbearing potential has a negative urine pregnancy test result and agrees to use a medically approved method of birth control. Acceptable methods of birth control include: hormonal contraceptives such as oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System); double-barrier methods; non-hormonal intrauterine devices; vasectomy of partner; and non-heterosexual lifestyles.
6. Subject agrees to discontinue the use of pre- and/or probiotic and/or polyphenol supplements from 30 days prior to the screening visit and throughout the study.
7. Subject agrees to consume less than 1/2 cup/day of foods containing anthocyanins (such as blueberries, blackberries, bilberries, cherries, grapes, grape juice, pomegranate, raspberries, huckleberries, strawberries) and no more than 1 glass/day of red wine, 3 cups/day of tea or coffee, or 10 g/day of dark chocolate from 30 days prior to the screening visit and throughout the study.
8. No known allergies to study products or components (bilberries, black currants, rice).
9. Subject is willing and able to completely consume high-fat meal and assigned study products within 15 min.
10. Subject is willing to consume a low fat/low flavonoid dinner the evening before visits 2, 3 and 5.
11. Subject has received a complete COVID-19 vaccine and is at least 6 weeks post-vaccine at the screening visit as verified by shot record or similar documentation.
12. Subject has given voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

1. Age < 18 or > 40 years.
2. BMI < 21 or > 29.9 kg/m2.
3. Vegan, Vegetarian, or other dietary restrictions that would not allow the subject to consume the high-fat meal.
4. Current consumption of special diets (e.g. Atkins, keto, paleo, etc.).
5. Current participation or enrollment in another pharmaceutical, weight-loss or nutritional clinical study within the last 30 days. Device trials are exempted.
6. Regular participation in endurance exercise activities (e.g. marathon running, triathlons).
7. Uncontrolled hypertension defined as diastolic blood pressure ≥ 95 mmHg and/or systolic blood pressure ≥ 160 mmHg.
8. Fasting blood triglycerides > 150 mg/dL.
9. Plasma amount of triglycerides accumulated in 5 h < 170 or > 700 mg/dL x 5 h after high-fat meal consumption at screening visit.
10. Self-reported Type 2 Diabetes
11. Fasting blood glucose < 50 mg/dL or > 100 mg/dL.
12. Hemoglobin A1c levels ≥ 5.7%.
13. Current smoker or use of tobacco products within the last 180 days.
14. Binge drinking (alcohol intake ≥ 5 alcoholic drinks for males or ≥ 4 alcoholic drinks for females on the same occasion, i.e. at the same time or within a couple of hours of each other).
15. Substance abuse or dependence within the last 60 days.
16. Daily use of anti-inflammatory medications including NSAIDs and aspirin within the last 30 days.
17. Use of laxative medications or other products that promote colon cleansing within the last 30 days.
18. History of restricted diets or use of herbal supplements or medications that interfere with insulin metabolism within the last 30 days.
19. History of stroke, hepatic, kidney, thyroid disease or cancer.
20. History of immune related disorders or Raynaud's disease.
21. Current clinically significant depression, anxiety or other psychiatric condition.
22. History of malabsorption or GI tract disorders.
23. History of GI surgeries (e.g. lap band, gastric bypass, etc.).
24. Diarrhea or oral antibiotic intake within the last 30 days.
25. Weight change (> 5%) within the last 30 days.
26. History of eating disorders such as bulimia, anorexia, or muscle dysmorphia.
27. Allergy or sensitivity to the study products or components of the high-fat meal.
28. Subject has not received a complete COVID-19 vaccine or is less than 6 weeks post-vaccine at the screening visit.
29. Any other condition which in the Investigator's opinion might adversely affect the subject's ability to complete the study or its measurements or which might pose significant risk to the subject.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in plasma triglycerides at week 8, both at fasting and at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to measure triglycerides in plasma

SECONDARY OUTCOMES:
Change from baseline in plasma free fatty acids at week 8, both at fasting and at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to measure plasma free fatty acids in plasma
Change from baseline in total free fatty acids at week 8, both at fasting and at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to measure total free fatty acids in plasma
Change from baseline in HDL at week 8, both at fasting and at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to measure HDL in plasma
Change from baseline in LDL at week 8, both at fasting and at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to measure LDL in plasma
Change from baseline in glucose at week 8, both at fasting and at week 8, both at fasting and at 0.25hr, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to measure glucose in plasma
Change from baseline in insulin at week 8, both at fasting and at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to measure insulin in plasma
Change from baseline in LPS at week 8, both at fasting and at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to measure LPS in plasma
Change from baseline in LPS binding protein at week 8, both at fasting and at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to measure LPS binding protein in plasma
Change from baseline in insulin resistance at week 8, both at fasting and at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to measure insulin resistance in PBMCs
Change from baseline in PBMC gene expression at week 8, both at fasting and at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to isolate RNA and measure gene expression in PBMCs. The most significantly differentially expressed transcripts will be chosen for further analysis.
Change from baseline in plasma total polyphenols at week 8, both at fasting and at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to measure total polyphenols in plasma
Change from baseline in plasma total anthocyanidins at week 8, both at fasting and at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to measure total anthycyanidins in plasma
Change from baseline in plasma Irisin at week 8, both at fasting and at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to measure Irisin in plasma
Change from baseline in total blood gene expression at week 8, both at fasting and at 3hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood sample collected by venipuncture to isolate RNA and measure gene expression in whole blood. The most significantly deferentially expressed transcripts will be chosen for further analysis.
Change from baseline in blood pressure at week 8, both at fasting and at 1hrs, 2hrs, 3hrs, 4hrs, and 5hrs post high-fat meal consumption | Baseline, 8 weeks
  blood pressure measured by sphygmomanometer
Change from baseline in fecal microbiota composition at week 8 | Baseline, 8 weeks
  stool sample collected to measure gut microbiota composition using 16S rRNA gene sequences
Change from baseline in fecal short chain fatty acids at week 8 | Baseline, 8 weeks
  stool sample collected to measure fecal short chain fatty acids
Change from baseline in skin carotenoids at week 4, and week 8 | baseline, 4 weeks, 8 weeks
  skin carotenoid scanner will be used to produce a raman score of skin carotenoids

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Oteiza, PhD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Nutrition Department, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Undecided